CLINICAL TRIAL: NCT01730820
Title: Influence of Preload Dependence on the Effect of Phenylephrine on Cardiac Output
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: NEO CO; A12-D20-VOL12 (Other: Basse Normandie FRANCE ethics committee)
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The perioperative hemodynamic management aims to ensure organ perfusion pressure and an oxygen arterial transport adapted to oxygen consumption. Phenylephrine is the α-adrenergic agonist widely used during anesthesia for arterial pressure control.

Several questions on phenylephrine global and regional hemodynamics effects remain unresolved.

The investigators assume that Phenylephrine may decrease cardiac output by increasing the afterload, while most likely could also make an increase or a stability of cardiac output by action on the venous return. The investigators propose an observational study assessing the influence of preload dependence, defined by the values of pulse pressure variation, on the effect of phenylephrine on cardiac output, measured beat by beat by esophageal Doppler.

The aim of the investigators work is to improve the understanding of phenylephrine action, a daily use therapeutic action, to improve the patients care.

ELIGIBILITY:
Inclusion Criteria:

* Hypotension (SBP <90 mm Hg and / or MAP <60 mm Hg)
* Injection of a bolus of phenylephrine at the discretion of the anesthesiologist physician in charge of the patient.

Exclusion Criteria:

* Minor or major patient under guardianship
* Esophageal Diseases
* supra ventricular rhythm trouble
* Severe valvular
* Shunt intracardiac
* Vt <7ml/kg theoretical weight
* heart rate / respiratory rate <3.6
* Clinical hypepression of intra-abdominal
* Compliance <30 mL/cmH2O
* pulmonary hypertension, Right ventricular failure
* Spontaneous Ventilation
* Thorax open
* VG severe dysfunction (LVEF <40%)
* Prior Injection of ephedrine prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General anesthesia.Orotracheal intubation and mechanical ventilation Advanced Hemodynamic Monitoring intraoperative ( arterial pressure catheter, esophageal Doppler)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
cardiac output | one year
  Comparing cardiac output values before and after injection of a phenylephrine bolus, based on the existence of a preload dependency, defined by a measure of respiratory variation of pulse pressure greater than or equal to 13%.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier REBET, M.D, Principal Investigator — University Hospital, Caen
Locations (1):
- CAEN University Hospital, Caen, Basse Normandie, France

REFERENCES:
- [Derived] Rebet O, Andremont O, Gerard JL, Fellahi JL, Hanouz JL, Fischer MO. Preload dependency determines the effects of phenylephrine on cardiac output in anaesthetised patients: A prospective observational study. Eur J Anaesthesiol. 2016 Sep;33(9):638-44. doi: 10.1097/EJA.0000000000000470. PMID 27164015